CLINICAL TRIAL: NCT04946942
Title: Implementing a Family Caregiver Checklist in Primary Care: A Pilot Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Weill Medical College of Cornell University (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: 21-04023513; 5K01AG061275 (NIH)
Record Dates: First submitted 2021-06-23; First posted 2021-07-01 (Actual); Results first posted 2025-07-03 (Actual); Last update posted 2025-07-03 (Actual); Status verified 2025-06

CONDITIONS: Caregiver Burnout
Keywords: Caregiver; Older adult; Primary care; Screening
MeSH Terms: conditions — Caregiver Burden | interventions — Caregivers

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Caregiver Checklist (CHEC) (Experimental): CHEC is composed of two elements: 1) a checklist to identify the needs and concerns of unpaid/family caregivers who accompany older adults (aged 65+) to their primary care visits and 2) Tip Sheet for clinicians.
  Interventions: Behavioral: Collaborative Healthcare Encounters with Caregivers (CHEC)
- Usual care (Active Comparator): Attendance at primary care appointments as usual.
  Interventions: Behavioral: Usual Care

INTERVENTIONS:
Behavioral: Collaborative Healthcare Encounters with Caregivers (CHEC) — CHEC is a brief checklist designed to identify family caregivers' unmet needs and concerns.
  Arms: Caregiver Checklist (CHEC)
Behavioral: Usual Care — Attendance at primary care appointments as usual.
  Arms: Usual care

SUMMARY:
The goal of this project is to pilot test CHEC (Collaborative Healthcare Encounters with Caregivers) in primary care. CHEC is brief intervention with two components: 1) a checklist to identify the needs and concerns of unpaid/family caregivers who accompany older patients (aged 65+) to their primary care visits and 2) accompanying Tip Sheet for clinicians.

ELIGIBILITY:
Inclusion Criteria:

Patients

* Age 65-89
* English speaking
* Women and men
* Of varying race/ethnicity
* Accompanied to primary care visits at the Center on Aging by a family caregiver (family caregiver also consents to participating in this study)
* Sufficient cognitive capacity to consent themselves or through a legal representative

Caregivers

* Age 21+
* English speaking
* Women and men
* Of varying race/ethnicity
* Accompany an older adult to his or her primary care visits at the Center on Aging (Older adult also consents to participating in this study)
* Cognitively intact (on basis of a 6-item cognitive screen)

Clinicians

* Age 21+
* Women and men
* Of varying race/ethnicity
* Treat patients at the Center on Aging

Exclusion Criteria:

* Patients, caregivers, and clinicians that do not meet the inclusion criteria.
* Patients and caregivers who are deaf or have hearing impairments that limit their ability to answer telephone queries.
* Caregivers who are visually impaired and cannot see well enough to read large print and complete paper-based surveys.
* Patients and/or caregivers whose dyad counterpart does not consent to take part in the study (i.e., Patients gives consent and their caregiver does not).

Ages: 21 Years to 89 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 113 (Actual)
Dates: Start 2021-08-30 (Actual); Primary Completion 2024-08-27 (Actual); Study Completion 2024-12-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Catherine Riffin, PhD, Principal Investigator — Weill Medical College of Cornell University; Karl Pillemer, PhD, Principal Investigator — Cornell University
Locations (1):
- Weill Cornell Medicine, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Neprash HT, Everhart A, McAlpine D, Smith LB, Sheridan B, Cross DA. Measuring Primary Care Exam Length Using Electronic Health Record Data. Med Care. 2021 Jan;59(1):62-66. doi: 10.1097/MLR.0000000000001450. PMID 33301282
- [Derived] Riffin C, Brody L, Wolff JL, Pillemer KA. A Pilot Trial Evaluating Collaborative Healthcare Encounters With Caregivers: A Checklist-Based Intervention for Primary Care. J Appl Gerontol. 2025 Dec;44(12):2006-2014. doi: 10.1177/07334648251323688. Epub 2025 Feb 27. PMID 40015556

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The trial was conducted at an academic affiliated geriatrics practice in New York City.
Pre-assignment Details: Participants included primary care physicians, patients, and their accompanying family caregivers. Physicians were were randomized 1:1 to CHEC or usual care using a computer-assisted algorithm to ensure unbiased allocation. Patient-caregiver dyads of participating physicians were allocated to CHEC or usual care based on the randomization of their assigned physician. The counts below for the CHEC and Usual Care arms include patients and caregivers.
Groups:
- Clinicians: Participating physicians of the patients
Period: Overall Study
Arm/Group | Caregiver Checklist (CHEC) | Usual Care | Clinicians
Started | 58 (29 patients and 29 caregivers) | 48 (24 patients and 24 caregivers) | 7
Completed | 52 (26 patients and 26 caregivers) | 46 (23 patients and 23 caregivers) | 7
Not Completed | 6 | 2 | 0
Not completed — Lost to Follow-up | 6 | 2 | 0

BASELINE CHARACTERISTICS:
Population: Age was not collected for the 7 primary care physicians.
Groups:
- Caregiver Checklist (CHEC): Caregivers; Caregiver Checklist (CHEC): Patient: CHEC is composed of two elements: 1) a checklist to identify the needs and concerns of unpaid/family caregivers who accompany older adults (aged 65+) to their primary care visits and 2) Tip Sheet for clinicians.
  Collaborative Healthcare Encounters with Caregivers (CHEC): CHEC is a brief checklist designed to identify family caregivers' unmet needs and concerns.
- Usual Care: Caregiver; Usual Care: Patient: Attendance at primary care appointments as usual.
  Usual Care: Attendance at primary care appointments as usual.
- Total: Total of all reporting groups
Arm/Group | Caregiver Checklist (CHEC): Caregivers | Caregiver Checklist (CHEC): Patient | Usual Care: Caregiver | Usual Care: Patient | Clinicians | Total
Number analyzed (Participants) | 29 | 29 | 24 | 24 | 7 | 113
Age, Continuous [Mean (Standard Deviation); unit: years] — Population: Age was not collected for the 7 primary care physicians.
  years
    number analyzed (Participants) | 29 | 29 | 24 | 24 | 0 | 106
    (all) | 65.4 (11.4) | 86.9 (8.1) | 61.7 (13.0) | 86.2 (5.4) |  | 75.3 (15.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 27 | 14 | 15 | 18 | 4 | 78
  Male | 2 | 15 | 9 | 6 | 3 | 35
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 2 | 2 | 0 | 0 | 7
  Not Hispanic or Latino | 26 | 23 | 21 | 20 | 7 | 97
  Unknown or Not Reported | 0 | 4 | 1 | 4 | 0 | 9
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 3 | 3 | 0 | 0 | 2 | 8
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 0 | 0 | 0 | 1
  Black or African American | 2 | 2 | 2 | 3 | 0 | 9
  White | 19 | 18 | 20 | 16 | 5 | 78
  More than one race | 3 | 5 | 1 | 3 | 0 | 12
  Unknown or Not Reported | 1 | 1 | 1 | 2 | 0 | 5
Region of Enrollment [Number; unit: participants]
  United States | 29 | 29 | 24 | 24 | 7 | 113

OUTCOME MEASURES:

1. Primary Outcome: The Number of Caregivers Who Complete the Checklist
Description: The number of caregivers who complete the checklist
Time Frame: Through study completion, up to 1 year
Population: Only caregivers assigned to the CHEC condition (n=28) were analyzed for this outcome measure. The patients from these dyads were not assessed for this measure.
Measure: Count of Participants; unit: Participants
Arm/Group | Caregiver Checklist (CHEC) | Usual Care
Number analyzed (Participants) | 28 | 0
Participants | 28 |

2. Primary Outcome: Acceptable Length of CHEC, as Measured by the Number of Caregivers Who Report That the Checklist is an Acceptable Length
Description: Acceptable length of CHEC, as measured by the number of caregivers who report that the checklist is an acceptable length
Time Frame: Post intervention, at 1 week
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Caregiver Checklist (CHEC) | Usual Care
Number analyzed (Participants) | 28 | 0
Participants | 23 |

3. Primary Outcome: CHEC's Ease of Use, as Measured by the Number of Caregivers Who Report That the Checklist is Easy to Use
Description: CHEC's ease of use, as measured by the number of caregivers who report that the checklist is easy to use
Time Frame: Post intervention, at 1 week
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Caregiver Checklist (CHEC) | Usual Care
Number analyzed (Participants) | 28 | 0
Participants | 25 |

4. Primary Outcome: CHEC's Helpfulness in Identify Caregivers' Needs, as Measured by the Number of Caregivers Who Report That the Checklist is Helpful in Identifying Their Needs
Description: CHEC's helpfulness in identify caregivers' needs, as measured by the number of caregivers who report that the checklist is helpful in identifying their needs
Time Frame: Post intervention, at 1 week
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Caregiver Checklist (CHEC) | Usual Care
Number analyzed (Participants) | 28 | 0
Participants | 20 |

5. Primary Outcome: CHEC's Helpfulness in Starting a Conversation With Health Care Providers About Caregivers' Needs, as Measured by the Number of Caregivers Who Report That the Checklist is Helpful in Starting a Conversation With Providers About Their Needs
Description: CHEC's helpfulness in starting a conversation with health care providers about caregivers' needs, as measured by the number of caregivers who report that the checklist is helpful in starting a conversation with providers about their needs
Time Frame: Post intervention, at 1 week
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Caregiver Checklist (CHEC) | Usual Care
Number analyzed (Participants) | 28 | 0
Participants | 22 |

6. Primary Outcome: Desire to Continue Use, as Measured by the Number Caregivers Who Report That They Desire to Continue Using the Checklist in the Future
Description: Desire to continue use, as measured by the number caregivers who report that they desire to continue using the checklist in the future
Time Frame: Post intervention, at 1 week
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Caregiver Checklist (CHEC) | Usual Care
Number analyzed (Participants) | 28 | 0
Participants | 15 |

7. Primary Outcome: Discussion of Caregivers' Needs, as Measured by the Number of Completed Checklists That Result in a Conversation With Providers About Caregiver Needs/Concerns
Description: Discussion of caregivers' needs, as measured by the number of completed checklists that result in a conversation with providers about caregiver needs/concerns
Time Frame: Post intervention, at 1 week
Population: as for outcome 1
Measure: Number; unit: checklists
Arm/Group | Caregiver Checklist (CHEC) | Usual Care
Number analyzed (Participants) | 28 | 0
checklists | 22 |

ADVERSE EVENTS:
Time Frame: 6 months
Description: Clinicians were not assessed for adverse events.
Groups:
- Caregiver Checklist (CHEC): Caregiver; Caregiver Checklist (CHEC): Patient: CHEC is composed of two elements: 1) a checklist to identify the needs and concerns of unpaid/family caregivers who accompany older adults (aged 65+) to their primary care visits and 2) Tip Sheet for clinicians.
  Collaborative Healthcare Encounters with Caregivers (CHEC): CHEC is a brief checklist designed to identify family caregivers' unmet needs and concerns.
Arm/Group | Caregiver Checklist (CHEC): Caregiver | Caregiver Checklist (CHEC): Patient | Usual Care: Caregiver | Usual Care: Patient
All-Cause Mortality (participants affected / at risk) | 0/29 | 0/29 | 0/24 | 0/24
Serious Adverse Events (participants affected / at risk) | 0/29 | 0/29 | 0/24 | 0/24
Other Adverse Events (participants affected / at risk) | 0/29 | 0/29 | 0/24 | 1/24
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Caregiver Checklist (CHEC): Caregiver (N=29) | Caregiver Checklist (CHEC): Patient (N=29) | Usual Care: Caregiver (N=24) | Usual Care: Patient (N=24)
Patient/care recipient abuse (Social circumstances) | 0 | 0 | 0 | 1

LIMITATIONS AND CAVEATS:
As a small feasibility trial, the study was not powered to conduct multivariable analyses that account for caregiver characteristics or to evaluate treatment effects by time. Additionally, findings may not generalize to mainstream primary care practice, given that recruitment occurred at a single academic geriatrics clinic with generous appointment lengths that may have enabled greater discussion of caregiver concerns.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-05-02): https://cdn.clinicaltrials.gov/large-docs/42/NCT04946942/Prot_SAP_000.pdf